CLINICAL TRIAL: NCT05159934
Title: Nicotine Discrimination in Smokers
Brief Title: Nicotine Differences in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: MS063
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Twenty participants will have 2 Experimental Session on 2 separate days. Experimental Session 1 will determine if smokers can reliably discriminate 0.1mg nicotine/pulse nicotine from saline. Experimental Session 2 will determine if smokers can discriminate 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine from saline.
Who Masked: Participant, Investigator
Masking Description: Nicotine dose will be prepared by pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine (Active Comparator): Experimental Session 2 will determine if smokers can discriminate 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine from saline.
  Interventions: Drug: Saline
- saline (Placebo Comparator): Saline will compared to different nicotine doses. Nicotine doses: 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine from saline.
  Interventions: Drug: 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine

INTERVENTIONS:
Drug: 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine — Determine if smokers can discriminate 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine from saline.
  Arms: saline
Drug: Saline — Saline will be use to determine if smokers can discriminate from the nicotine/pulse of nicotine and saline
  Arms: Nicotine

SUMMARY:
The primary aim of this project is to determine the threshold dose of nicotine, which the smokers will be able to differentiate from placebo (saline). Will use IV pulsed-nicotine infusion that closely matches nicotine delivery by inhaled tobacco use (i.e., tobacco cigarette or electronic cigarette), allowing precise and reproducible nicotine delivery. Four nicotine doses (0.1, 0.05, 0.025, and 0.0125 mg nicotine/pulse) which are within the range of nicotine doses that are delivered by cigarettes with very low to regular nicotine content. These doses will be delivered as a cluster of 4 pulsed-nicotine infusions of 2 sec duration with a 28 sec interval between each dose.

DETAILED DESCRIPTION:
Twenty participants will have 2 Experimental Session on 2 separate days. Experimental Session 1 will determine if smokers can reliably discriminate 0.1mg nicotine/pulse nicotine from saline. Experimental Session 2 will determine if smokers can discriminate 0.05, 0.025, and 0.0125 mg nicotine/pulse of nicotine from saline.

Hypothesis: The threshold for discrimination will be 0.05 mg nicotine/pulse and the doses below that (0.025, and 0.0125 mg nicotine/pulse) will be subthreshold.

Exploratory Aim: To explore the relationship between the threshold for subjective drug effects and drug discrimination.

ELIGIBILITY:
Inclusion criteria:

* Female and male smokers, aged 18 to 65 years veterans and non-veterans who have been smoking tobacco cigarettes for at least a year
* smoke ≥ 5 cigs/day ;
* urine cotinine levels > 100 ng/mL consistent with nicotine intake of an active smoker (23)
* not seeking treatment at the time of the study for nicotine dependence
* Good health as verified by medical history, screening examination, and screening laboratory tests
* For women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion criteria:

* History of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the subject to be in the study
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* current alcohol or substance dependence for any other recreational or prescription drugs other than nicotine
* use of e-cigarettes more than 10 days in the past 30 days
* urine drug screening indicating recent illicit drugs use (with the exception of marijuana).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Drug Effect Questionnaire | over 3 hours
  Liking effect

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States